CLINICAL TRIAL: NCT03108833
Title: A Phase IIa Trial to Assess the Efficacy and Safety of Recombinant Human Prourokinase in the Treatment of Acute Pulmonary Embolism
Brief Title: A Trial in Recombinant Human Prourokinase to Treat Acute Pulmonary Embolism
Acronym: ERUPTE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tasly Biopharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TASLY-B1448
Record Dates: First submitted 2017-04-05; First posted 2017-04-11 (Actual); Last update posted 2021-03-18 (Actual); Status verified 2021-03

CONDITIONS: Acute Pulmonary Embolism
MeSH Terms: interventions — Tissue Plasminogen Activator

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Low Dose Experimental Group (Experimental): Recombinant Human Prourokinase:40mg
  Interventions: Drug: Recombinant Human Prourokinase
- High Dose Experimental Group (Experimental): Recombinant Human Prourokinase:50mg
  Interventions: Drug: Recombinant Human Prourokinase
- Active Comparator Controlled Group (Active Comparator): Alteplase:100mg if weight>=65kg, 1.5mg/kg if weight<65kg
  Interventions: Drug: Alteplase

INTERVENTIONS:
Drug: Recombinant Human Prourokinase — The drug is used for intravenous thrombolysis therapy
  Other Names: rhPro-UK
  Arms: High Dose Experimental Group; Low Dose Experimental Group
Drug: Alteplase — The drug is used for intravenous thrombolysis therapy
  Other Names: Actilyse; rtPA
  Arms: Active Comparator Controlled Group

SUMMARY:
This trial is being conducted to assess the efficacy and safety of recombinant Human Prourokinase in the acute pulmonary embolism.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-75 years（Include the critical value）AND
2. High-risk PE or medium high-risk PE AND
3. PE symptom duration ≤14 days AND
4. PLT≥100×10^9/L，ALT and AST≤2.5ULN，TBIL<ULN，Cr within the normal range AND
5. Informed consent can be obtained from subject or Legally Authorized Representative

Exclusion Criteria:

1. Hemorrhagic or unexplained stroke history
2. Ischemic stroke or transient ischemic attack (TIA) within 6 months
3. The existence of the central nervous system injury or tumor
4. Severe trauma，major surgery or head injury within 3 weeks
5. Active bleeding within 1 month
6. Clinician deems high-risk for bleeding
7. Using anticoagulants (after a washout period can be randomized)
8. Pregnancy or delivery within 1 week
9. Vascular puncture which can not be oppressed
10. Cardiopulmonary resuscitation within 10 days
11. Systolic blood pressure above 180 mmHg or diastolic blood pressure above 100mmHg
12. Severe liver dysfunction
13. Infective endocarditis
14. Arterial aneurysm or arteriovenous malformation or suspected aortic dissection
15. left atrial thrombus
16. Neurosurgery or eye surgery within 1 month
17. Hemorrhagic diabetic retinopathy
18. Serious cardiac insufficiency
19. ventricular arrhythmias
20. Known allergic to prourokinase，urokinase，recombinant tissue-type plasminogen activator，contrast agent or any drug in the trial
21. Do not allow for 30 days' study
22. Any disease or condition is not suitable for intravenous thrombolysis
23. Lactating women or plan to pregnant women during the trial，or don't want to during the study period using effective contraception or abstinence of male and female patients with possibility of fertility
24. Clinician thinks patient doesn't fit to participate in the test of other diseases or conditions

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2017-06-06 (Actual); Primary Completion 2019-12-19 (Actual); Study Completion 2019-12-19 (Actual)

PRIMARY OUTCOMES:
Qanadli CT Score | 0 and 48hours after treatment
  Change of Qanadli Score from baseline by CTPA 48hours after treatment
Average pulmonary artery pressure | 0,24hours，48hours，7days and 30days after treatment
  Changes of average pulmonary artery pressure from baseline 24hours，48hours，7days and 30days after treatment
Three tricuspid regurgitation velocity | 0,24hours，48hours，7days and 30days after treatment
  Changes of Three tricuspid regurgitation velocity from baseline 24hours，48hours，7days and 30days after treatment
RV to LV Diameter Ratio(Ultrasonic echocardiography) | 0,24hours，48hours，7days and 30days after treatment
  Changes of RV to LV Diameter Ratio from baseline 24hours，48hours，7days and 30days after treatment
RV to LV Diameter Ratio(CTPA) | 0,24hours，48hours，7days and 30days after treatment
  Changes of RV to LV Diameter Ratio from baseline 24hours，48hours，7days and 30days after treatment
Pulmonary systolic pressure | 0,24hours，48hours，7days and 30days after treatment
  Changes of pulmonary systolic pressure from baseline 24hours，48hours，7days and 30days after treatment
NT-proBNP | 0，48hours and 30days after treatment
  Changes of NT-proBNP from baseline 48hours and 30days after treatment
Major bleeding | From baseline to 30 days
  The frequency of major bleeding
bleeding | From baseline to 30 days
  The frequency of bleeding
Incidence of death from all causes | From baseline to 7 days
  Incidence of death from all causes
Incidence of recurrent pulmonary embolism | From baseline to 7 days
  Incidence of recurrent pulmonary embolism
Incidence of death from all causes | From baseline to 30 days
  Incidence of death from all causes
Incidence of hemodynamic deterioration | From baseline to 7 days
  Incidence of hemodynamic deterioration

CONTACTS AND LOCATIONS:
Locations (18):
- China (18):
  - Fuwai Hospital, Beijing, Beijing Municipality
  - Anzhen Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Beijing Tongren Hospital,Capital Medical University, Beijing, Beijing Municipality
  - The Second Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang
  - Henan Provincial People's Hospital, Zhengzhou, Henan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Wuhan Asia Heart Hospital, Wuhan, Hubei
  - Xiangya Hospital, Central South University, Changsha, Hunan
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - Nanjing First Hospital, Nanjing, Jiangsu
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - The First Hospital of Jilin University, Changchun, Jilin
  - The First Hospital of China Medical University, Shenyang, Liaoning
  - General Hospital of Ningxia Medical University, Yinchuan, Ningxia
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi’an, Shanxi
  - West China Hospital of Sichuan University, Chengdu, Sichuan
  - Tianjin Chest Hospital, Tianjin, Tianjin Municipality
  - Sir Run Run Shaw Hospital affiliated with the Zhejiang University School of Medicine, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No